CLINICAL TRIAL: NCT03813550
Title: Intestinal Microbiota and Vitamin K Levels in PXE Patients (IMPROVE Study)
Acronym: IMPROVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Maastricht University (Other); Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018/79
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: PXE; calcification; Gla proteins; gut microbiota; vitamin K2; menaquinones; taxonomic meta-sequencing
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Calcinosis | interventions — Defecation; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PXE cohort 2019-2020 (Other): PXE patient cohort monitored at referral centre from 2019 to 2020: fecal and blood samples
  Interventions: Diagnostic Test: Fecal and blood samples

INTERVENTIONS:
Diagnostic Test: Fecal and blood samples — Fecal samples for intestinal microbiota analysis; Blood and fecal samples for assessment of various forms of vitamin K

SUMMARY:
This study aims to demonstrate a potential association between gut microbiota composition, plasma levels of various forms of vitamin K, and severity of clinical manifestations of Pseudoxanthoma Elasticum (PXE).

DETAILED DESCRIPTION:
Vitamin K deficiency contributes to pathological calcification which underlies the clinical picture of pseudoxanthoma elasticum (PXE), an inherited autosomal recessive disease. A substantial proportion of vitamin K, namely the K2 form (menaquinones), is produced by gut microbiota. In healthy volunteers fecal levels of the major menaquinone producers, Escherichia coli and Bacteroides species, are approximately 5 and 9 log10 CFU/g dry weight respectively. There is however a lack of data on gut microbiota in PXE patients. The objective of our project is to demonstrate a potential association between gut microbiota composition, plasma levels of various forms of vitamin K and severity of clinical manifestations in PXE patients.

This study will be performed as Research surrounding bio collection "Clinical and biological exploration of PXE patients" kept at the Center of Biological Resources of Angers University Hospital (bio collection n° DC 20116-14-67, authorization to transfer n° 2016-27-99). Fecal samples, plasma samples and clinical data will be collected from patients diagnosed with PXE who will be monitored at the Angers University Hospital Referral Center (France) in 2019-2020. Clinical severity of PXE will be assessed using modified Phenodex score. Gut microbiota will be analyzed using metagenomic sequencing. Plasma Vitamin K species and fecal excretion of menaquinones will be assessed using HPLC. Plasma dp-ucMGP (circulating biomarker of vitamin K status) and serum PIVKA-II (protein induced by vitamin K absence-II) will be assessed using immunoassay. Results will be compared to healthy age- and gender-matched controls from the pre-existing Biofortis database.

ELIGIBILITY:
Inclusion Criteria:

* Patients with phenotypically and genetically (ABCC6) proven PXE
* Aged over 18 years
* Written consent obtained for Angers University Hospital (France) PXE bio-collection

Exclusion Criteria:

* Patients under the age of 18
* Patients unwilling to participate in the study, or unable to sign the bio-collection consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Fecal samples for intestinal microbiota analysis | 15 min
  Gut microbiota composition and relative abundance of species (via metagenomic sequencing)
Fecal samples for assessment of various forms of vitamin K | 15 min
  Fecal Vitamin K species
Blood samples for assessment of various forms of vitamin K | 15 min
  Plasma Vitamin K species
Blood samples for assessment of dp-ucMGP | 15 min
  Plasma dp-ucMGP
Blood samples for assessment of PIVKA-II | 15 min
  Serum PIVKA-II
Severity of ocular and cardiovascular PXE manifestations and extent of PXE skin changes | 15 min
  Modified Phenodex score:
  * Skin lesions severity: S0=No sign; S1= Papules/bumps; S2= Plaques of coalesced papules; S3= Lax and redundant skin
  * Number of affected skin sites: for Typical and Nontypical areas
  * Ophthalmological involvement: E0= No sign; E1= Peau d'orange ; E2= Angioid streaks; E3a=Medical history of bleeding and/or scarring; E3b= Unilateral or bilateral blindness
  * Gastrointestinal bleeding: G0= No sign; G1= Gastrointestinal bleeding as related to PXE
  * Vascular involvement: V0= No sign; V1= Weak or absent pulse or peripheral artery disease revealed by vascular imaging; V2= Intermittent claudication; V3= Medical history of vascular surgery or Stroke/TIA
  * Cardiac involvement: C0= No sign; C1= medical history of chest pain/angina/abnormal EKG or abnormal stress test with no symptom, or Mitral insufficiency; C2= Heart attack
  * Renal involvement: R0= No sign; R1a= asymptomatic nephrocalcinosis revealed by imaging; R1b= Nephrolithiasis

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic MARTIN, MD, PhD, Principal Investigator — Department of Dermatology, University Hospital of Angers
Locations (3):
- France (2):
  - Biofortis Mérieux NutriSciences, Saint-Herblain, Pays de la Loire Region
  - Department of Dermatology, University Hospital of Angers, Angers, Pays de Loire
- Department of Biochemistry, University Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jansen RS, Duijst S, Mahakena S, Sommer D, Szeri F, Varadi A, Plomp A, Bergen AA, Oude Elferink RP, Borst P, van de Wetering K. ABCC6-mediated ATP secretion by the liver is the main source of the mineralization inhibitor inorganic pyrophosphate in the systemic circulation-brief report. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):1985-9. doi: 10.1161/ATVBAHA.114.304017. Epub 2014 Jun 26. PMID 24969777
- [Background] Jansen RS, Kucukosmanoglu A, de Haas M, Sapthu S, Otero JA, Hegman IE, Bergen AA, Gorgels TG, Borst P, van de Wetering K. ABCC6 prevents ectopic mineralization seen in pseudoxanthoma elasticum by inducing cellular nucleotide release. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20206-11. doi: 10.1073/pnas.1319582110. Epub 2013 Nov 25. PMID 24277820
- [Background] Pomozi V, Brampton C, van de Wetering K, Zoll J, Calio B, Pham K, Owens JB, Marh J, Moisyadi S, Varadi A, Martin L, Bauer C, Erdmann J, Aherrahrou Z, Le Saux O. Pyrophosphate Supplementation Prevents Chronic and Acute Calcification in ABCC6-Deficient Mice. Am J Pathol. 2017 Jun;187(6):1258-1272. doi: 10.1016/j.ajpath.2017.02.009. Epub 2017 Apr 14. PMID 28416300
- [Background] Gheduzzi D, Boraldi F, Annovi G, DeVincenzi CP, Schurgers LJ, Vermeer C, Quaglino D, Ronchetti IP. Matrix Gla protein is involved in elastic fiber calcification in the dermis of pseudoxanthoma elasticum patients. Lab Invest. 2007 Oct;87(10):998-1008. doi: 10.1038/labinvest.3700667. Epub 2007 Aug 27. PMID 17724449
- [Background] Hendig D, Zarbock R, Szliska C, Kleesiek K, Gotting C. The local calcification inhibitor matrix Gla protein in pseudoxanthoma elasticum. Clin Biochem. 2008 Apr;41(6):407-12. doi: 10.1016/j.clinbiochem.2007.12.023. Epub 2008 Jan 11. PMID 18222176
- [Background] Li Q, Jiang Q, Schurgers LJ, Uitto J. Pseudoxanthoma elasticum: reduced gamma-glutamyl carboxylation of matrix gla protein in a mouse model (Abcc6-/-). Biochem Biophys Res Commun. 2007 Dec 14;364(2):208-13. doi: 10.1016/j.bbrc.2007.09.122. Epub 2007 Oct 4. PMID 17942075
- [Background] Vanakker OM, Martin L, Schurgers LJ, Quaglino D, Costrop L, Vermeer C, Pasquali-Ronchetti I, Coucke PJ, De Paepe A. Low serum vitamin K in PXE results in defective carboxylation of mineralization inhibitors similar to the GGCX mutations in the PXE-like syndrome. Lab Invest. 2010 Jun;90(6):895-905. doi: 10.1038/labinvest.2010.68. Epub 2010 Apr 5. PMID 20368697
- [Background] Gorgels TG, Waarsing JH, Herfs M, Versteeg D, Schoensiegel F, Sato T, Schlingemann RO, Ivandic B, Vermeer C, Schurgers LJ, Bergen AA. Vitamin K supplementation increases vitamin K tissue levels but fails to counteract ectopic calcification in a mouse model for pseudoxanthoma elasticum. J Mol Med (Berl). 2011 Nov;89(11):1125-35. doi: 10.1007/s00109-011-0782-y. Epub 2011 Jul 2. PMID 21725681
- [Background] Shearer MJ, Bach A, Kohlmeier M. Chemistry, nutritional sources, tissue distribution and metabolism of vitamin K with special reference to bone health. J Nutr. 1996 Apr;126(4 Suppl):1181S-6S. doi: 10.1093/jn/126.suppl_4.1181S. PMID 8642453
- [Background] Ramotar K, Conly JM, Chubb H, Louie TJ. Production of menaquinones by intestinal anaerobes. J Infect Dis. 1984 Aug;150(2):213-8. doi: 10.1093/infdis/150.2.213. PMID 6470528
- [Background] Shearer MJ. Vitamin K. Lancet. 1995 Jan 28;345(8944):229-34. doi: 10.1016/s0140-6736(95)90227-9. No abstract available. PMID 7823718
- [Background] Walther B, Karl JP, Booth SL, Boyaval P. Menaquinones, bacteria, and the food supply: the relevance of dairy and fermented food products to vitamin K requirements. Adv Nutr. 2013 Jul 1;4(4):463-73. doi: 10.3945/an.113.003855. PMID 23858094
- [Background] Bentley R, Meganathan R. Biosynthesis of vitamin K (menaquinone) in bacteria. Microbiol Rev. 1982 Sep;46(3):241-80. doi: 10.1128/mr.46.3.241-280.1982. No abstract available. PMID 6127606
- [Background] Conly JM, Stein K. The production of menaquinones (vitamin K2) by intestinal bacteria and their role in maintaining coagulation homeostasis. Prog Food Nutr Sci. 1992 Oct-Dec;16(4):307-43. PMID 1492156
- [Background] Beulens JW, Booth SL, van den Heuvel EG, Stoecklin E, Baka A, Vermeer C. The role of menaquinones (vitamin K(2)) in human health. Br J Nutr. 2013 Oct;110(8):1357-68. doi: 10.1017/S0007114513001013. Epub 2013 Apr 16. PMID 23590754
- [Background] Conly JM, Stein K. Quantitative and qualitative measurements of K vitamins in human intestinal contents. Am J Gastroenterol. 1992 Mar;87(3):311-6. PMID 1539565
- [Background] Schurgers LJ, Teunissen KJ, Hamulyak K, Knapen MH, Vik H, Vermeer C. Vitamin K-containing dietary supplements: comparison of synthetic vitamin K1 and natto-derived menaquinone-7. Blood. 2007 Apr 15;109(8):3279-83. doi: 10.1182/blood-2006-08-040709. Epub 2006 Dec 7. PMID 17158229
- [Background] Suttie JW. The importance of menaquinones in human nutrition. Annu Rev Nutr. 1995;15:399-417. doi: 10.1146/annurev.nu.15.070195.002151. PMID 8527227
- [Background] Usui Y, Tanimura H, Nishimura N, Kobayashi N, Okanoue T, Ozawa K. Vitamin K concentrations in the plasma and liver of surgical patients. Am J Clin Nutr. 1990 May;51(5):846-52. doi: 10.1093/ajcn/51.5.846. PMID 2333843
- [Background] Berkner KL, Runge KW. The physiology of vitamin K nutriture and vitamin K-dependent protein function in atherosclerosis. J Thromb Haemost. 2004 Dec;2(12):2118-32. doi: 10.1111/j.1538-7836.2004.00968.x. PMID 15613016
- [Background] Cranenburg EC, Schurgers LJ, Vermeer C. Vitamin K: the coagulation vitamin that became omnipotent. Thromb Haemost. 2007 Jul;98(1):120-5. PMID 17598002
- [Background] McCann JC, Ames BN. Vitamin K, an example of triage theory: is micronutrient inadequacy linked to diseases of aging? Am J Clin Nutr. 2009 Oct;90(4):889-907. doi: 10.3945/ajcn.2009.27930. Epub 2009 Aug 19. PMID 19692494
- [Background] Shearer MJ. Role of vitamin K and Gla proteins in the pathophysiology of osteoporosis and vascular calcification. Curr Opin Clin Nutr Metab Care. 2000 Nov;3(6):433-8. doi: 10.1097/00075197-200011000-00004. PMID 11085828
- [Background] Shanahan CM, Proudfoot D, Farzaneh-Far A, Weissberg PL. The role of Gla proteins in vascular calcification. Crit Rev Eukaryot Gene Expr. 1998;8(3-4):357-75. doi: 10.1615/critreveukargeneexpr.v8.i3-4.60. PMID 9807700
- [Background] Schurgers LJ, Spronk HM, Soute BA, Schiffers PM, DeMey JG, Vermeer C. Regression of warfarin-induced medial elastocalcinosis by high intake of vitamin K in rats. Blood. 2007 Apr 1;109(7):2823-31. doi: 10.1182/blood-2006-07-035345. PMID 17138823
- [Background] Li Q, Guo H, Chou DW, Harrington DJ, Schurgers LJ, Terry SF, Uitto J. Warfarin accelerates ectopic mineralization in Abcc6(-/-) mice: clinical relevance to pseudoxanthoma elasticum. Am J Pathol. 2013 Apr;182(4):1139-50. doi: 10.1016/j.ajpath.2012.12.037. Epub 2013 Feb 15. PMID 23415960
- [Background] Luo G, Ducy P, McKee MD, Pinero GJ, Loyer E, Behringer RR, Karsenty G. Spontaneous calcification of arteries and cartilage in mice lacking matrix GLA protein. Nature. 1997 Mar 6;386(6620):78-81. doi: 10.1038/386078a0. PMID 9052783
- [Background] Theuwissen E, Smit E, Vermeer C. The role of vitamin K in soft-tissue calcification. Adv Nutr. 2012 Mar 1;3(2):166-73. doi: 10.3945/an.111.001628. PMID 22516724
- [Background] Shea MK, O'Donnell CJ, Hoffmann U, Dallal GE, Dawson-Hughes B, Ordovas JM, Price PA, Williamson MK, Booth SL. Vitamin K supplementation and progression of coronary artery calcium in older men and women. Am J Clin Nutr. 2009 Jun;89(6):1799-807. doi: 10.3945/ajcn.2008.27338. Epub 2009 Apr 22. PMID 19386744
- [Background] Vermeer C, Shearer MJ, Zittermann A, Bolton-Smith C, Szulc P, Hodges S, Walter P, Rambeck W, Stocklin E, Weber P. Beyond deficiency: potential benefits of increased intakes of vitamin K for bone and vascular health. Eur J Nutr. 2004 Dec;43(6):325-35. doi: 10.1007/s00394-004-0480-4. Epub 2004 Feb 5. PMID 15309455
- [Background] Geleijnse JM, Vermeer C, Grobbee DE, Schurgers LJ, Knapen MH, van der Meer IM, Hofman A, Witteman JC. Dietary intake of menaquinone is associated with a reduced risk of coronary heart disease: the Rotterdam Study. J Nutr. 2004 Nov;134(11):3100-5. doi: 10.1093/jn/134.11.3100. PMID 15514282
- [Background] Gast GC, de Roos NM, Sluijs I, Bots ML, Beulens JW, Geleijnse JM, Witteman JC, Grobbee DE, Peeters PH, van der Schouw YT. A high menaquinone intake reduces the incidence of coronary heart disease. Nutr Metab Cardiovasc Dis. 2009 Sep;19(7):504-10. doi: 10.1016/j.numecd.2008.10.004. Epub 2009 Jan 28. PMID 19179058
- [Background] Beulens JW, Bots ML, Atsma F, Bartelink ML, Prokop M, Geleijnse JM, Witteman JC, Grobbee DE, van der Schouw YT. High dietary menaquinone intake is associated with reduced coronary calcification. Atherosclerosis. 2009 Apr;203(2):489-93. doi: 10.1016/j.atherosclerosis.2008.07.010. Epub 2008 Jul 19. PMID 18722618
- [Background] Brandenburg VM, Schurgers LJ, Kaesler N, Pusche K, van Gorp RH, Leftheriotis G, Reinartz S, Koos R, Kruger T. Prevention of vasculopathy by vitamin K supplementation: can we turn fiction into fact? Atherosclerosis. 2015 May;240(1):10-6. doi: 10.1016/j.atherosclerosis.2015.02.040. Epub 2015 Feb 24. PMID 25744701
- [Background] Caluwe R, Pyfferoen L, De Boeck K, De Vriese AS. The effects of vitamin K supplementation and vitamin K antagonists on progression of vascular calcification: ongoing randomized controlled trials. Clin Kidney J. 2016 Apr;9(2):273-9. doi: 10.1093/ckj/sfv146. Epub 2015 Dec 29. PMID 26985380
- [Background] Jandhyala SM, Talukdar R, Subramanyam C, Vuyyuru H, Sasikala M, Nageshwar Reddy D. Role of the normal gut microbiota. World J Gastroenterol. 2015 Aug 7;21(29):8787-803. doi: 10.3748/wjg.v21.i29.8787. PMID 26269668
- [Background] Carrillo-Linares JL, Garcia-Fernandez MI, Morillo MJ, Sanchez P, Rioja J, Baron FJ, Ariza MJ, Harrington DJ, Card D, Boraldi F, Quaglino D, Valdivielso P. The Effects of Parenteral K1 Administration in Pseudoxanthoma Elasticum Patients Versus Controls. A Pilot Study. Front Med (Lausanne). 2018 Apr 16;5:86. doi: 10.3389/fmed.2018.00086. eCollection 2018. PMID 29713628
- [Background] Brampton C, Yamaguchi Y, Vanakker O, Van Laer L, Chen LH, Thakore M, De Paepe A, Pomozi V, Szabo PT, Martin L, Varadi A, Le Saux O. Vitamin K does not prevent soft tissue mineralization in a mouse model of pseudoxanthoma elasticum. Cell Cycle. 2011 Jun 1;10(11):1810-20. doi: 10.4161/cc.10.11.15681. Epub 2011 Jun 1. PMID 21597330
- [Background] Karlsson FH, Fak F, Nookaew I, Tremaroli V, Fagerberg B, Petranovic D, Backhed F, Nielsen J. Symptomatic atherosclerosis is associated with an altered gut metagenome. Nat Commun. 2012;3:1245. doi: 10.1038/ncomms2266. PMID 23212374